CLINICAL TRIAL: NCT07266675
Title: Post-Acute Phase of Cardiogenic Shock (PACS) Registry
Brief Title: Post-Acute Phase of Cardiogenic Shock
Status: Recruiting | Type: Observational
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 24MMHIS216e
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-10

CONDITIONS: Cardiogenic Shock
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Epidemiology studies showed that the burden of cardiogenic shock (CS) persistently high, with increasing annual medical expenses and steady prevalence. In-hospital and one-year mortality reduce annually. Hence, there are increasing number of patients who survive to hospital discharge but they will face further challenges in the subacute stage after hospital discharge. However, there are still insufficient studies focusing on this issue. Establishment of a healthcare neatwork to help hospital survivors of CS return society safely is critical.

DETAILED DESCRIPTION:
Multicener, prospective cohort study

ELIGIBILITY:
Inclusion Criteria:

Hospital survivors of cardiogenic shock

Exclusion Criteria:

* Age < 18 years。
* Patient or family refuse follow-up.
* Patient died within hospital stay.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital survivors of cardiogenic shock
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
mortality | 1 year
  any death
rehospitalization | 1 year
  any rehospitalization

SECONDARY OUTCOMES:
mortality | 90-day
  any death
rehospitalization | 90-day
  any rehospitalization
mortality | 180-day
  any death
rehospitalization | 180-day
  any rehospitalization

OTHER OUTCOMES:
Quality | 1 year
  KCCQ

CONTACTS AND LOCATIONS:
Overall Officials: Cardiovascular department, Principal Investigator — Mackay Memorial Hospital
Locations (1):
- MacKay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
need further discussion with other PI

REFERENCES:
- [Background] Chien SC, Hsu CY, Liu HY, Lin CF, Hung CL, Huang CY, Chien LN. Cardiogenic shock in Taiwan from 2003 to 2017 (CSiT-15 study). Crit Care. 2021 Nov 18;25(1):402. doi: 10.1186/s13054-021-03820-1. PMID 34794502
- [Background] Shah M, Patil S, Patel B, Agarwal M, Davila CD, Garg L, Agrawal S, Kapur NK, Jorde UP. Causes and Predictors of 30-Day Readmission in Patients With Acute Myocardial Infarction and Cardiogenic Shock. Circ Heart Fail. 2018 Apr;11(4):e004310. doi: 10.1161/CIRCHEARTFAILURE.117.004310. PMID 29618581
- [Background] Vallabhajosyula S, Payne SR, Jentzer JC, Sangaralingham LR, Kashani K, Shah ND, Prasad A, Dunlay SM. Use of Post-Acute Care Services and Readmissions After Acute Myocardial Infarction Complicated by Cardiac Arrest and Cardiogenic Shock. Mayo Clin Proc Innov Qual Outcomes. 2021 Feb 8;5(2):320-329. doi: 10.1016/j.mayocpiqo.2020.12.006. eCollection 2021 Apr. PMID 33997631
- [Background] Shah M, Patnaik S, Patel B, Ram P, Garg L, Agarwal M, Agrawal S, Arora S, Patel N, Wald J, Jorde UP. Trends in mechanical circulatory support use and hospital mortality among patients with acute myocardial infarction and non-infarction related cardiogenic shock in the United States. Clin Res Cardiol. 2018 Apr;107(4):287-303. doi: 10.1007/s00392-017-1182-2. Epub 2017 Nov 13. PMID 29134345
- [Background] Shah RU, de Lemos JA, Wang TY, Chen AY, Thomas L, Sutton NR, Fang JC, Scirica BM, Henry TD, Granger CB. Post-Hospital Outcomes of Patients With Acute Myocardial Infarction With Cardiogenic Shock: Findings From the NCDR. J Am Coll Cardiol. 2016 Feb 23;67(7):739-47. doi: 10.1016/j.jacc.2015.11.048. PMID 26892407
- [Background] Aissaoui N, Puymirat E, Simon T, Bonnefoy-Cudraz E, Angoulvant D, Schiele F, Benamer H, Quandalle P, Prunier F, Durand E, Berard L, Blanchard D, Danchin N. Long-term outcome in early survivors of cardiogenic shock at the acute stage of myocardial infarction: a landmark analysis from the French registry of Acute ST-elevation and non-ST-elevation Myocardial Infarction (FAST-MI) Registry. Crit Care. 2014 Sep 19;18(5):516. doi: 10.1186/s13054-014-0516-y. PMID 25246084
- [Background] Chien SC, Wang CA, Liu HY, Lin CF, Huang CY, Chien LN. Comparison of the prognosis among in-hospital survivors of cardiogenic shock based on etiology: AMI and Non-AMI. Ann Intensive Care. 2024 May 12;14(1):74. doi: 10.1186/s13613-024-01305-2. PMID 38735891